CLINICAL TRIAL: NCT03319264
Title: Sarcopenia in Axial and Peripheral Spondyloarthropathies
Acronym: SASPAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 69HCL17_0145; 2017-A02391-52 (Other: ID-RCB)
Record Dates: First submitted 2017-10-18; First posted 2017-10-24 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Spondylarthropathy; Sarcopenia
Keywords: Spondylarthropathy; Sarcopenia; lean mass; fat mass
MeSH Terms: conditions — Spondylarthropathies; Sarcopenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with SpA (Experimental): Patients included in this single group study will have 3 interventions to assess the severity of muscle loss :
  * dynamometry exam
  * walking test
  * Dual-energy X-ray Absorptiometry (DXA) measurement Quality of life will be assessed with Sarcopenia & Quality of Life (SARQOL) questionnaire. Patients will also fill a Life habits Questionnaire.
  Interventions: Other: Dynamometry exam; Other: Walking test; Radiation: DXA measurement; Other: SARQOL questionnaire; Behavioral: Life habits Questionnaire

INTERVENTIONS:
Other: Dynamometry exam — Prehension strength of the main hand will be assessed thanks to dynamometry, in order to evaluate patient's muscular strength
Other: Walking test — A 4 metres walking test will be performed to assess patient's walking speed
Radiation: DXA measurement — DXA measurement will be performed to assess patient's body composition
Other: SARQOL questionnaire — Patient's quality of life will be assessed thanks to the SARQOL questionnaire
Behavioral: Life habits Questionnaire — Life habits Questionnaire

SUMMARY:
Spondylarthropathies (SpA) are among the most common chronic inflammatory rheumatisms in adults, responsible for a muscular loss or sarcopenia which can be very disabling, not much documented in the literature, and not yet studied in France. In addition, sarcopenia is associated with decreased physical activity and increased risk of falls and fractures. A better characterization of the determinants of this muscular loss will allow to better detect and take care of it.

The aim is to conduct the first French study on the prevalence and severity of sarcopenia in patients with spondyloarthropathies and to study the variables that may be associated with it. Finally, we propose to evaluate obesity related to sarcopenia in these patients and compare them to cases matched for age and sex (from OFELY / STRAMBO cohorts, Lyon, FRANCE).

This is a prospective interventional and monocentric study with minimal risks and constraints: patients will be included for one day for an evaluation of their sarcopenia by measuring their muscle strength, physical performance and body composition and recording of their socio-demographic and disease characteristics.

ELIGIBILITY:
Inclusion Criteria:

* Men and women, 18 to 80 years old
* Hospitalized or attending the rheumatology department for spondyloarthopathy.

Exclusion Criteria:

* no signed consent
* Immobilization for a period of more than 15 days during the last 3 months
* pregnant or breastfeeding woman
* Not affiliated to the national healthcare insurance
* difficulty in understanding French
* psychiatric disorder

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2017-11-02 (Actual); Primary Completion 2018-07-04 (Actual); Study Completion 2018-07-04 (Actual)

PRIMARY OUTCOMES:
Muscular strength | At day 1
  Muscular strength is the first outcome to evaluate sarcopenia
Walking speed | At day 1
  Walking speed is a physical performance outcome, that is the second outcome to evaluate sarcopenia
Muscular mass | Up to 4 month after inclusion
  Muscular mass is the third outcome to evaluate sarcopenia and will be assessed using DXA

SECONDARY OUTCOMES:
Alcohol consumption | At day 1
Tobacco consumption | At day 1
Time of sport practice per month | At day 1
  Number of hours of sport practice per month is the first outcome to evaluate patient's global physical activity.
Physical activity rate in work | At day 1
  Physical activity rate in work can be light, medium, high or not applicable if the patient does not work ; it is the second outcome to evaluate patient's physical global activity.
Average walking time in a week | At day 1
  Average walking time in a week is the third outcome to evaluate patient's physical global activity.
Score at the SARQOL questionnaire | At day 1
  Quality of life will be assessed thanks to the SARQOL questionnaire (score between 0 and 100)

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Rhumatologie - Hôpital Edouard Herriot, Lyon, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Merle B, Cottard M, Sornay-Rendu E, Szulc P, Chapurlat R. Spondyloarthritis and Sarcopenia: Prevalence of Probable Sarcopenia and its Impact on Disease Burden: The Saspar Study. Calcif Tissue Int. 2023 Jun;112(6):647-655. doi: 10.1007/s00223-023-01074-3. Epub 2023 Mar 21. PMID 36944706